CLINICAL TRIAL: NCT01907763
Title: A 12-week, Multi-center, Randomized, Double Blinded, Parallel Group, Placebo-controlled Study to Assess the Efficacy and Safety of SOTB07 in Asthma Patients
Brief Title: Study Phase III Study to Assess the Efficacy and Safety of SOTB07 in Asthma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOTB07_AST_III_2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: asthma; SOTB07
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SOTB07 200mg (Experimental): One tablet of SOTB07 200mg and One tablet of SOTB 400mg Placebo are administered twice a day.
  Interventions: Drug: SOTB07 200mg; Drug: SOTB 400mg placebo
- SOTB07 400mg (Experimental): One tablet of SOTB07 400mg and One tablet of SOTB 200mg Placebo are administered twice a day.
  Interventions: Drug: SOTB07 400mg; Drug: SOTB 200mg placebo
- Placebo (Placebo Comparator): One tablet of SOTB 200mg Placebo and One tablet of SOTB 400mg Placebo are administered twice a day.
  Interventions: Drug: SOTB 200mg placebo; Drug: SOTB 400mg placebo

INTERVENTIONS:
Drug: SOTB07 200mg
  Arms: SOTB07 200mg
Drug: SOTB07 400mg
  Arms: SOTB07 400mg
Drug: SOTB 200mg placebo — Placebo of SOTB07 200mg
  Arms: Placebo; SOTB07 400mg
Drug: SOTB 400mg placebo — Placebo of SOTB07 400mg
  Arms: Placebo; SOTB07 200mg

SUMMARY:
The objective of this study is to assess the efficacy and safety of SOTB07 in asthma patients by observing changes FEV1 (% predicted) as the primary efficacy endpoint after oral administration of SOTB07 200mg, 400mg, placebo for 12 weeks.

DETAILED DESCRIPTION:
A 12-week, Multi-center, Randomized, Double blinded, Parallel group, Placebo-controlled study to Assess the Efficacy and Safety of SOTB07 in asthma patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or eligible female subjects aged 15 years or more
2. A female is eligible if she is of:

   * Non-child bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is at least 2 year after post- menopausal
   * Child bearing potential and agrees to the acceptable contraceptive methods used consistently and correctly
   * Negative pregnancy test at screening
3. Non-smoker for at least 1 year, a pack history of ≤ 10 pack years
4. Symptom of persistent asthma, as defined by the National Institute of Health (NIH) 5.50% ≤ FEV1 ≤ 80% predicted at screening visit (withholding inhaled, short acting ß-agonist for 6 hours)

6.FEV1 reversibility ≥ 12% and 200 ml at 20-30 minutes after inhalation of a short acting ß-agonist (Salbutamol 2 puffs; 200㎍) at Visit 1 or within 6 months before Visit 1 7.Capable of withholding salbutamol use for ≥ 6 hours prior to clinic visits 8.Appropriately signed and dated informed consent has been obtained

Exclusion Criteria:

1. Active upper or lower respiratory tract infection within 3 weeks before visit 1
2. Emergency room treatment for asthma within 1 month or hospitalization for asthma within 3 months before visit 1
3. Any evidence of infectious, oncologic, or other active pulmonary disease obtained by chest radiography within 12 months before visit 1
4. Clinically significant, in the opinion of the investigator, hematological, liver, renal, heart, neurological disease, or other serious disease
5. Hypersensitivity to any β2-agonist, sympathomimetic drug, leukotriene receptor antagonist or Sophora tonkinensis Radix Rhizoma
6. Clinically significant and uncontrolled psychiatric disease
7. history of drug or alcohol abuse
8. Inhaled, oral or parenteral corticosteroids within 4 weeks before visit 1
9. Change of Immunotherapy within 6 months before visit 1
10. Administration of the antiasthma agent within 1 week of visit 1
11. Administration of any other medication which may affect the course of asthma, or interact with sympathomimetic amines
12. Participation in study using an experimental medication within 1 month before visit 1
13. Other ineligible subject in the opinion of the investigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
FEV1 change from the baseline | 12 weeks

SECONDARY OUTCOMES:
Change in spirometer parameters | 12 weeks
Change in FeNO | 12 weeks
Change in AM/PM PEFR | 12 weeks
Change in diurnal asthma symptom score | 12 weeks
Change in the number of days with experience of nocturnal asthma symptoms | 12 weeks
Change in amount of beta-2 agonist used (puff/day) | 12 weeks
Proportion of rescue free day | 12 weeks
Proportion of asthma control day | 12 weeks
Proportion of asthma exacerbation | 12 weeks
Proportion of treatment failure (severe asthma exacerbation) | 12 weeks
Changes in asthma control questionaire score | 12 weeks
Changes in quality of life questionaire for adult korea asthmatics scores | 12 weeks
Changes in patient's global self assessment score | 12 weeks
Change in visual analogue scale for cough score | 12 weeks
Change in biomarkers (eosinophil, neutrophil, ECP, eotaxin) in blood sample | 12 weeks
Change in biomarkers (eosinophil, neutrophil, ECP, eotaxin) in sputum sample | 12 weeks
Assessment of Safety | 12 weeks
  Adverse Event/ Vital Sign/ Laboratory Test

CONTACTS AND LOCATIONS:
Overall Officials: Sangheon Cho, professor, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea